CLINICAL TRIAL: NCT01520168
Title: The 2005 Composix Kugel Mesh Recall Leaves Unresolved Problems of Patient Management: Taking Stock After 5-year Follow up
Brief Title: Composix Kugel Mesh Recall Leaves Unresolved Problems of Patient Management
Status: Suspended | Type: Observational
Why Stopped: Because of the product recall 2005/2006.
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, PD Dr. Dr. Ulrich A. Dietz, PD Dr. Dr., University of Wuerzburg
Other Study IDs: UD 069/11
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; Mesh; Surgery; Composix Kugel; IPOM technique
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Explanted meshes
Oversight: Data Monitoring Committee: No

SUMMARY:
From its introduction in 2000 until its US recall in December 2005, the Composix Kugel Mesh was implanted in an estimated 350,000 patients worldwide.

The purpose of the study is to evaluate retrospectively the complications related to this mesh that occurred in our patients between 2003 and 2005, since new complications continue to be diagnosed, although the investigators discontinued the use of the mesh.

DETAILED DESCRIPTION:
From 2003 to 2005(2006) we implanted Komposix Kugel Meshes in 21 Patients with incisional ventral hernias. With the recall of January 2006 (in Germany), we stopped the implantation of this mesh and continued to monitor the patients with follow up and phone interviews. Late complications still continue to occur, mainly as a consequence of the product defect identified 7 years ago.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Incisional hernia

Exclusion Criteria:

* Younger than 18 years
* Peritonitis
* Intestinal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) with the diagnosis of symptomatic incisional hernia.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2003-10; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Early postoperative complications | 6 months postoperative
  Assessment of postoperative complications (wound complication, mesh infection, seroma)

SECONDARY OUTCOMES:
Long-term postoperative complications | 6 months to 5 years
  Chronic pain, chronic and recurrent mesh infection, mesh bulging, incisional hernia and intestinal fistula

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich A. Dietz, MD, PhD, Principal Investigator — University of Wuerzburg
Locations (1):
- Department of General, Visceral, Vascular and Pediatric Surgery, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Muysoms FE, Bontinck J, Pletinckx P. Complications of mesh devices for intraperitoneal umbilical hernia repair: a word of caution. Hernia. 2011 Aug;15(4):463-8. doi: 10.1007/s10029-010-0692-x. Epub 2010 Jun 17. PMID 20556448
- [Background] LeBlanc KA, Whitaker JM. Management of chronic postoperative pain following incisional hernia repair with Composix mesh: a report of two cases. Hernia. 2002 Dec;6(4):194-7. doi: 10.1007/s10029-002-0075-z. Epub 2002 Sep 11. PMID 12424601
- [Background] Hope WW, Iannitti DA. An algorithm for managing patients who have Composix Kugel ventral hernia mesh. Hernia. 2009 Oct;13(5):475-9. doi: 10.1007/s10029-009-0498-x. Epub 2009 Apr 4. PMID 19347564
- [Background] Robinson TN, Clarke JH, Schoen J, Walsh MD. Major mesh-related complications following hernia repair: events reported to the Food and Drug Administration. Surg Endosc. 2005 Dec;19(12):1556-60. doi: 10.1007/s00464-005-0120-y. Epub 2005 Oct 5. PMID 16211441
- [Background] Dietz UA, Spor L, Germer CT. [Management of mesh-related infections]. Chirurg. 2011 Mar;82(3):208-17. doi: 10.1007/s00104-010-2013-4. German. PMID 21327906
- See also: Research page of the Department — http://www.zom-wuerzburg.de/index.php?id=236